CLINICAL TRIAL: NCT07005414
Title: Efficacy of Bumetanide in Children With Autism Spectrum Disorder Guided by Peripheral Blood Biomarkers and Machine Learning Models: A Randomized Controlled Trial
Brief Title: Efficacy of Bumetanide in Children With Autism Spectrum Disorder Guided by Peripheral Blood Biomarkers and Machine Learning Models
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fei Li (Other)
Responsible Party: Sponsor-Investigator, Fei Li, Chief Physician, Doctoral Supervisor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XHEC-C-2025-089
Record Dates: First submitted 2025-05-25; First posted 2025-06-05 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Bumetanide; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bumetanide plus treatment as usual (TAU) (Experimental): Participants in experimental group will receive bumetanide, along with treatments as usual (i.e. behavioral interventions)
  Interventions: Drug: Bumetanide; Behavioral: Treatment as usual (TAU)
- Treatment as usual (TAU) (Other): Participants will undergo treatment as usual, such as behavioral interventions
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Drug: Bumetanide — Participants will receive bumetanide (0.5mg bid) for a period of three months.
  Arms: bumetanide plus treatment as usual (TAU)
Behavioral: Treatment as usual (TAU) — Participants will undergo treatment as usual, such as behavioral interventions

SUMMARY:
The objective of this study is to learn if bumetanide could alleviate the clinical symptoms in children with autism spectrum disorder (ASD), who has been predicted as high responders to bumetanide via a cytokine-based predictive model. The Eligible ASD participants identified as high responder to bumetanide will be randomly assigned to either the experimental group or the control group. Participants in the experimental group will receive bumetanide interventions, along with the behavioral interventions, for three months. Participants in the control group will only undergo behavioral interventions. The clinical symptoms and potential adverse effects will be closely monitored throughout the intervention period.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) affects about 1% children around the world and can cause lifelong disability and elevate premature mortality. Currently, no medication that can cure ASD or its core symptoms. The recent success of repurposing drugs for novel treatments in psychiatry has been highlighted, with one of the examples given being the use of bumetanide to improve the core symptoms in ASD. However, the heterogeneity in the treatment effect of bumetanide among ASD patients has been observed. A further study (Li et al., Translational Psychiatry, 2022) demonstrated that integrating the cytokine levels and behavioral symptoms could help to identify optimal responders to bumetanide in ASD, showing promise for biomarker- and machine learning model-guided precision medicine with bumetanide.

This open-label clinical trial aimed at investigating whether bumetanide could alleviate the clinical symptoms in children with ASD predicted as high responders to bumetanide via a cytokine-based predictive model. The Eligible ASD participants identified as high responder to bumetanide will be randomly assigned to either the experimental group or the control group. Participants in the experimental group will receive bumetanide interventions, along with the behavioral interventions, for a period of three months. Participants in the control group will only undergo behavioral interventions. The clinical symptoms and potential adverse effects will be closely monitored throughout the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 3 and 6 years old
* Meeting the ASD diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* Meeting the ASD diagnostic criteria of the Diagnostic Observational Scale for Autism, Second Edition(ADOS-2)
* CARS total score ≥ 30
* Identified as high responder to bumetanide by machine learning algorithms
* Obtaining informed consent from the legal guardian

Exclusion Criteria:

* Liver and kidney dysfunction
* With a history of allergy to sulfa drugs
* History of neurological diseases such as epilepsy
* Abnormal ECG
* Diagnosed with genetic or chromosomal abnormalities
* Brain structural abnormalities detected by MRI which required surgical intervention
* Using the melatonin treatment for sleep disorders or withdrawal less than three weeks.
* Received any new intervention within 8 weeks prior to enrollment

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Social Responsiveness Scale, Second Edition (SRS-2) | From enrollment to the end of treatment at 3 months
  Social Responsiveness Scale, Second Edition (SRS-2) is a scale used to evaluate the presence and severity of social impairment. The scores of the SRS-2 rate from 0 to 195, and higher scores indicate more severe symptoms. Changes of the SRS-2 scores from baseline to 3 month after treatment will be analyzed to assess the effect of the intervention on children with ASD.

SECONDARY OUTCOMES:
Clinical Global Impressions Scale (CGI) | From enrollment to the end of treatment at 3 months
  Clinical Global Impressions Scale (CGI) is a scale used to assess the severity of the illness and the global improvement of the participants under intervention.The Clinical Global Impression - Severity scale (CGI-S) is a clinician rated 7-point measure of overall severity. Scores range from 1 (Normal, not at all ill) through 4 (Moderately ill) to 7 (Among the most extremely ill patients). The Clinical Global Impression - Improvement scale (CGI-I) is the companion measure that evaluates the change in the patient's symptoms relative to baseline. Scores range from 1 (Very much improved) through 4 (No Change) to 7 (Very much worse).
Vineland Adaptive Behavior Scale | From enrollment to the end of treatment at 3 months
  The VABS is used to measure adaptive functioning across domains such as communication, daily living skills, socialization, and motor skills. Changes in VABS scores from baseline to 3 months post-treatment will be analyzed to assess the intervention's impact on adaptive behaviors in children with ASD.
Childhood Autism Rating Scale (CARS) | From enrollment to the end of treatment at 3 months
  CARS is a behavior-rating scale used to assess the presence and severity of the symptoms associated autism spectrum disorder. The scores of the CARS rate from 15 to 60, and higher scores indicate more severe symptoms. The changes in the CARS scores from baseline to 3 months after the treatment will be analyzed to assess the impact of the intervention on participants with ASD.
Aberrant Behavior Checklist (ABC) | From enrollment to the end of treatment at 3 months
  Aberrant Behavior Checklist (ABC) is a 58-item instrument used to measure behavior problems across five sub-scales: hyperactivity, irritability, social withdrawal, stereotypic behavior and inappropriate speech. Each item rates behavior severity on a 4 point scale from 0 (Not at all a problem) to 3 (The problem is severe in degree). A higher score indicates more frequent aberrant behaviors.Changes of the total scores and scores of subscales from baseline to 3 month after treatment will be analyzed.
Chinese Communicative Development Inventory (CCDI) | From enrollment to the end of treatment at 3 months
  Chinese Communicative Development Inventory (CCDI) is a questionnaire used to measures the language abilities. Higher scores suggest better language level. The changes in the CCDI between baseline and 3 month after treatment will be analyzed.

OTHER OUTCOMES:
Biomarkers (single nucleotide polymorphisms) | From enrollment to the end of treatment at 3 months
  Blood samples will be collected at baseline. Depending on funding availability, whole genome sequencing may subsequently be performed. If sequencing is conducted, a genome-wide association study will be carried out to investigate potential correlations between genetic polymorphisms and response to bumetanide treatment.
Biomarkers (metabolites) | From enrollment to the end of treatment at 3 months
  Blood samples will be collected at baseline and at the 3-month follow-up. Depending on funding availability, targeted metabolomics may subsequently be performed, covering free fatty acids, bile acids and amino acids profiling. Changes in the levels of metabolites between baseline and 3 months after treatment will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The Study Protocol, Statistical Analysis Plan, Informed Consent Form, and other relevant documents will be available under reasonable and ethically approved request to the corresponding authors.